CLINICAL TRIAL: NCT06112275
Title: WAYFINDER: A Clinical Study to Evaluate the Safety and Efficacy of ETX101, an AAV9-Delivered Gene Therapy in Children With SCN1A-positive Dravet Syndrome
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of ETX101, an AAV9-Delivered Gene Therapy in Children With SCN1A-positive Dravet Syndrome (Australia Only)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Encoded Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ETX-DS-004
Record Dates: First submitted 2023-10-25; First posted 2023-11-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-09

CONDITIONS: Dravet Syndrome
Keywords: Dravet; SCN1A; DEE; developmental and epileptic encephalopathy; Dravet Syndrome; SCN1A-positive; SCN1A+
MeSH Terms: conditions — Epilepsies, Myoclonic; Generalized Epilepsy With Febrile Seizures Plus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): Cohort A will evaluate ETX101 dose level 1.
  Interventions: Drug: ETX101
- Cohort B (Experimental): Cohort B will evaluate ETX101 dose level 2.
  Interventions: Drug: ETX101
- Cohort C (Experimental): Cohort C will evaluate ETX101 dose level 3.
  Interventions: Drug: ETX101
- Cohort D (Experimental): Cohort D will evaluate ETX101 dose level 4.
  Interventions: Drug: ETX101

INTERVENTIONS:
Drug: ETX101 — ETX101 is composed of a non-replicating, recombinant adeno-associated viral serotype 9 (rAAV9) vector used to deliver a GABAergic regulatory element (reGABA) and an engineered transcription factor that increases transcription of the SCN1A gene (eTFSCN1A).

SUMMARY:
WAYFINDER is a Phase 1/2 study in Australia to evaluate the safety and efficacy of ETX101 in participants with SCN1A-positive Dravet syndrome aged 6 to <84 months. The study follows an open-label, dose-escalation design.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a predicted loss of function pathogenic or likely pathogenic SCN1A variant.
* Participant must have experienced their first seizure between the ages of 3 and 15 months.
* Participant must have a clinical diagnosis of Dravet syndrome or the treating clinician must have a high clinical suspicion of a diagnosis of Dravet syndrome.
* Participant is receiving at least one prophylactic antiseizure medication.

Exclusion Criteria:

* Participant has another genetic mutation or clinical comorbidity which could potentially confound the typical Dravet phenotype.
* Participant has a known central nervous system structural and/or vascular abnormality (indicated by an MRI or CT scan of the brain).
* Participant has an abnormality that may interfere with CSF distribution and/or has an existing ventriculoperitoneal shunt.
* Participant is currently taking or has taken antiseizure medications (ASMs) at a therapeutic dose that are contraindicated in Dravet syndrome, including sodium channel blockers.
* Participant has experienced seizure freedom for a period of 4 consecutive weeks within the 6-month period prior to informed consent.
* Participant has previously received gene or cell therapy.
* Participant is currently enrolled in a clinical trial or receiving an investigational therapy.
* Participant has clinically significant underlying liver disease.

Ages: 6 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing any treatment-emergent adverse events (AEs), serious adverse events (SAEs), related AEs, AEs with severity Grade ≥ 3, AEs resulting in study discontinuation, and AEs with a fatal outcome. | Day 1 through Study Completion, an average of 5 years
Percent change from Baseline in monthly countable seizure frequency (MCSF) at Week 52, with countable seizures defined as generalized tonic-clonic/clonic, focal motor with clearly observable clinical signs, tonic bilateral, and atonic seizures. | Between the 8-week baseline period and the 48-week post-dosing assessment period (defined as Week 5 to Week 52 following administration of ETX101)
Proportion of participants free from episodes of prolonged seizures and/or status epilepticus at Week 52. | Week 5 through Week 52

SECONDARY OUTCOMES:
Proportion of participants with ≥ 90% reduction in monthly countable seizure frequency (MCSF) from Baseline at Week 52. | Between the 8-week baseline period and the 48-week post-dosing assessment period (defined as Week 5 to Week 52 following administration of ETX101)
Change from Baseline in the Vineland-Third Edition Expressive Communication raw score at Week 52. | Baseline through Week 52. Higher scores correspond to better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Rico, M.D., Ph.D, Study Director — Encoded Therapeutics
Locations (1):
- The Royal Children's Hospital, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No